CLINICAL TRIAL: NCT00547833
Title: Partial Word Knowledge Growth in Children With LLD
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1011841; 1R03DC006827-01A1 (NIH)
Record Dates: First submitted 2007-10-17; First posted 2007-10-23 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Language Disorders
Keywords: language disorders; language learning disabilities; vocabulary; reading
MeSH Terms: conditions — Language Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Experimental: Children with language-learning disabilities reading at approximately a 6th grade level
- Age-Matched: Typical language learners each of whom is pair match to an experimental participant by age and gender.
- Language-Matched: Typical language learners, each of whom is pair-matched to an experimental participant by reading comprehension skills and gender.

SUMMARY:
Children with language-learning disabilities (LLD) have language and reading skills that are weaker than those of typically developing children. In the school-age years, reading is a primary means of exposure to new vocabulary for typically developing children. Although these children would not be expected to master a new word through a single exposure to it in text, children show evidence of partial word knowledge growth (e.g., Wagovich & Newhoff, 2004). The purpose of this project is to characterize the partial word knowledge growth of children with LLD, in comparison to children with typical language skills. Five forms of partial word knowledge (e.g., orthographic, word discrimination, syntactic, emotional content, and general semantic domain knowledge) are being measured. The study's hypotheses are that children with LLD, like typically developing peers, will demonstrate partial word knowledge growth from exposure to unfamiliar words in text, but that they will show a different pattern of growth across the five forms of partial word knowledge being assessed.

DETAILED DESCRIPTION:
The purpose of this line of research is to examine the process by which children acquire partial meanings of unfamiliar words when they encounter the words for the first time in reading.

The proposed pilot study requires 6th grade children to attend three, 1-hour sessions, 2-3 days apart. The protocol for the present study is as follows: In the first session, the parents of the children will complete a consent form and a parent questionnaire; the children will complete an assent form, similar to the consent but with simpler language. Next, one half of the children will complete two pre-tests: a checklist and a multiple choice test; the other half will complete the checklist and a distracter task. In the second session, the children will read 2 of 4 possible stories, grade-appropriate in reading level and content. After reading each story, the children will be asked to write a one-page summary of the story. In the third session the children will all complete the checklist and multiple choice measure. These measures, as post-tests, are designed to assess the types of word knowledge children accrue when they read an unfamiliar word in a story.

The purpose of the proposed pilot study, then, is to assess the adequacy of the multiple choice measure, which is newly developed, for word knowledge measurement. In addition, the study will assess whether the group who received the multiple choice measure before reading the stories performs better on the posttests than the children who received only the checklist in the pretest phase. In sum, then, the purposes of the pilot are (a) to assess the adequacy of the new multiple choice measure for detecting word knowledge, and (b) to assess the adequacy of the design, prior to conducting the large-scale experiment later.

ELIGIBILITY:
Inclusion Criteria:

* test scores indicating language and/or reading difficulties
* reading at approximately a 6th grade level
* nonverbal cognitive screening within normal limits
* hearing screening within normal limits

Exclusion Criteria:

* history of neurological conditions such as seizure disorder or TBI
* history of emotional/behavior disorder

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Percent words learned for each of 5 partial word knowledge types | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stacy A Wagovich, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Univ. of Missouri Dept. of Communication Science & Disorders, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No